CLINICAL TRIAL: NCT06424093
Title: Effect of Virtual Reality Technology for Managment of Acute Pain in Outpatient Hysteroscopy: A Randomised Controlled Trial
Brief Title: Effect of Virtual Reality Technology for Managment of Acute Pain in Outpatient Hysteroscopy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Egymedicalpedia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Virtual Reality Technology
Record Dates: First submitted 2024-05-11; First posted 2024-05-21 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Acute Pain; Anxiety
Keywords: hysteroscopy; Acute Pain; Anxiety; Virtual Reality
MeSH Terms: conditions — Acute Pain; Anxiety Disorders | interventions — Hysteroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Cases Group (Experimental): About 25 women indicated for diagnostic hysteroscopy with using Virtual Reality Technology
  Interventions: Procedure: Virtual Reality Technology
- Group B: Control Group (Placebo Comparator): About 25 women indicated for diagnostic hysteroscopy without using Virtual Reality Technology
  Interventions: Procedure: Virtual Reality Technology

INTERVENTIONS:
Procedure: Virtual Reality Technology — To evaluate the role of virtual reality technology as distraction technique in the management of acute pain during outpatient hysteroscopy
  Other Names: Hysteroscopy

SUMMARY:
Performing out patient diagnostic and operative gynecological procedures is becoming more popular having the benefits of reducing risks of general anaesthetia, decreasing healthcare burden and increasing satisfaction for both patient and provider.

Virtual reality (VR), a new technology, has been studied as a distraction technique for non-pharmacological method of pain relief. It is a computer-generated representation of an immersive videos viewed through a headset.

DETAILED DESCRIPTION:
Performing out patient diagnostic and operative gynecological procedures is becoming more popular having the benefits of reducing risks of general anaesthetia, decreasing healthcare burden and increasing satisfaction for both patient and provider. Such procedures are usually well tolerated , However it can be associated with acute pain and anxiety. Options of Pain relief include sedation, local anaesthetic , analgesics and distraction techniques, however no consistent good quality evidence exists to support practice.

Virtual reality (VR), a new technology, has been studied as a distraction technique for non-pharmacological method of pain relief. It is a computer-generated representation of an immersive videos viewed through a headset. The obstacles of cost, quality and accessibility of (VR) devices have significantly eliminated in recent years and offer promising application in the medical field. Virtual reality for managing pain has been studied in many fields including paediatrics, dentistry, burns treatment, chronic pain, labour, and episiotomy.

Although a meta-analysis suggested that VR may have a role in reducing pain scores in acutely painful interventions , studies found it to be effective only in needles and burns physical therapy.

The studies of VR on pain and anxiety, however, were limited by clinical and statistical heterogeneity.

Nonpharmacological options of pain relief have not explored enough the role of VR in reducing pain and improving patient experience in outpatient hysteroscopy .To our knowledge, there is only one publication studying the role of virtual reality in the management of acute pain during office gynaecological procedures

ELIGIBILITY:
Inclusion Criteria:

- Patients scheduled for diagnostic hysteroscopy e.g. Infertility, AUB

Exclusion Criteria:

* Absolute contraindication to office hysteroscopy such as acute pelvic infection , active genital herpes , heavy bleeding or pregnancy.
* Psychological ,hearing or visual disorders.
* known anatomical condition that make performing office hysteroscopy is difficult such as cervical stenosis ,fibrosis or cervical amputation .
* Previous history of failed office hysteroscopy
* Patients scheduled for operative hysteroscopy.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-11-15 (Estimated)

PRIMARY OUTCOMES:
Assessment of Pain | 10 minutes from starting the procedure
  The pain level of the cases is evaluated by means of the digital pain as the 11-point visual analog scale (VAS) whereas 0-Represents no pain, 10 - Worst imaginable pain), as well as the 11-point VAS-A (0-Represents no anxiety, 10 - Highest anxiety)

CONTACTS AND LOCATIONS:
Overall Officials: Amr Elhussieny, Professor, Study Chair — Head of Obstetrics and Gynecology department , Faculty of Medicine, Ain Shams University; Mortada El Sayed Ahmed, Professor, Study Director — Department of obstetrics & gynecology, Faculty Of Medicine, Ain Shams University; Radwa Rsaheedy Ali, M.D, Principal Investigator — Department of obstetrics & gynecology, Faculty Of Medicine, Ain Shams University
Locations (1):
- Ain Shams University Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided